CLINICAL TRIAL: NCT05552638
Title: Feasibility to Embed Telecare in Rural Community Senior Centers
Brief Title: Telecare in Rural Senior Centers
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants enrolled into open trial during enrollment period.
Sponsor: Elizabeth K Rhodus (Other)
Responsible Party: Sponsor-Investigator, Elizabeth K Rhodus, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 78017
Record Dates: First submitted 2022-09-20; First posted 2022-09-23 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Health Care Utilization
Keywords: telehealth; rural; brain; aging
MeSH Terms: conditions — Patient Acceptance of Health Care | interventions — Telemedicine

STUDY DESIGN:
Intervention Model Description: Pre/Post-test design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Senior Center Members (Experimental): Participants who are using the provided telehealth stations in senior centers.
  Interventions: Other: Telecare

INTERVENTIONS:
Other: Telecare — The University of Kentucky (UK) will embed telehealth stations at community-based senior centers. Individuals who utilize these telehealth stations will be invited to complete a demographic survey prior to their telehealth appointment. Following their appointment, they will be invited to complete a semi-structured interview with the research team. Participants who elect to use telehealth station will be doing so as telehealth visits already scheduled with patients as Standard of Care (SOC). The telehealth station in the senior center will be used to increase ease and access to telehealth should the patient/provider choose to use such an approach (for example, in instances when the patient does not have sufficient technology, internet access, or capability to operate telehealth at home).

SUMMARY:
The objective of this project is to assess the feasibility of telehealth stations at community centers as a mechanism to increase healthcare access for older adults living in rural communities.

ELIGIBILITY:
Inclusion Criteria:

* Age of 21 years or older
* Independently capable to complete electronic survey form
* Cognitive capable to verbalize consent for semi-structured interview

Exclusion Criteria

- Unable to complete an electronic survey form

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-11-20 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of embedded telehealth stations in senior centers as mechanism to increase healthcare access for older adults. | 12 months
  Feasibility will be measured based on acceptance of the telehealth program by community residents evident by 5 Telehealth healthcare contacts per month

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No